CLINICAL TRIAL: NCT01727518
Title: The Austrian LEAD (Lung hEart sociAl boDy) Study
Acronym: LEAD
Status: Active, not recruiting | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Lung Health (Other)
Responsible Party: Sponsor
Other Study IDs: LEAD1
Record Dates: First submitted 2012-11-04; First posted 2012-11-16 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Respiration Disorders; Body Composition, Beneficial; Metabolic Health
Keywords: natural history; lung function; general population; metabolic health
MeSH Terms: conditions — Respiration Disorders; Glucocorticoid Receptor Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of urine and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reference Population: No Intervention
  Interventions: Other: As the LEAD study is an observational cohort study, there is no intervention to report.

INTERVENTIONS:
Other: As the LEAD study is an observational cohort study, there is no intervention to report. — As the LEAD study is an observational cohort study, there is no intervention to report.

SUMMARY:
The LEAD study is the first longitudinal cohort investigating respiratory, cardiac, and metabolic health in a reference population of Austria.

DETAILED DESCRIPTION:
The LEAD (Lung, hEart, sociAl, boDy) study is a longitudinal, observational, population-based cohort study aimed at investigating the prevalence and incidence of health disorders and the relationships between social, environmental, developmental, and aging factors that influence respiratory, cardiac, and metabolic health and comorbidities throughout life.

A random sample (male and female, age 6 - 80 years) of Vienna inhabitants (urban cohort) and all the inhabitants of six villages from Lower Austria (rural cohort) were invited to participate. Participants are followed up every four years. A number of investigations and measurements are obtained in each of the four domains of the study (Lung, hEart, sociAl, boDy), as briefly discussed below.

Lung Domain: Lung function measures include pre- and post-bronchodilation spirometry and static lung volumes, effort-independent measures of oscillatory resistance, and carbon monoxide lung diffusing capacity (DLCO). Measurements are obtained according to international recommendations, and reference values correspond to those of the Global Lung Function Initiative (GLI). Smoking history and exposure to environmental tobacco smoke (ETS) are recorded. History of respiratory diseases, allergies, and related medications from the individual and spouses, as well as respiratory symptoms, are collected using a questionnaire.

Heart Domain: Cardiovascular measurements include arterial blood pressure, automated electrocardiogram, carotid-femoral pulse wave velocity, and blood pressure measurements at both the upper and lower extremities. History of cardiovascular diseases and events, as well as related medications, are collected using a questionnaire.

Social Domain: Socioeconomic status (income, education, occupation) of the individual or parents/legal representative (if underage) is collected. To study the presence of neuropsychiatric diseases such as anxiety, depression, and impaired cognitive function, standardized questionnaires and test modules are used.

Body Domain: To determine the presence of diabetes and metabolic syndrome, we measure fasting glucose in peripheral venous blood, glycated hemoglobin (HbA1c), body mass index, waist circumference, fat mass, fat-free mass, blood lipid profiles, and blood pressure. The presence of osteoporosis is determined using dual-energy X-ray absorptiometry. History of diabetes, metabolic syndrome, and osteoporosis, as well as related medications from the individual, are collected using a questionnaire.

Blood and urine samples are analyzed for routine clinical measurements and stored in a biobank for future investigations.

All measurements are performed at the LEAD study center of the Ludwig Boltzmann Institute for Lung Health at the Otto Wagner Hospital in Vienna, Austria.

This health examination will be the first investigation in Austria providing information about the respiratory, cardiovascular, and metabolic health and relevant comorbidities in a longitudinal approach.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female,
* Age 6 - 80 years,
* Invitation by study invitation letter

Exclusion Criteria:

* Insufficient language skills
* pregnancy

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community based cohort
Sampling Method: Probability Sample
Enrollment: 14966 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2028-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robab Breyer-Kohansal, Prof. Dr., Principal Investigator — Ludwig Boltzmann Institute for Lung Health, Vienna, Austria; Marie-Kathrin Breyer, Prof. Dr, Study Director — Ludwig Boltzmann Institute for Lung Health, Vienna, Austria
Locations (1):
- The LEAD Study Center, Vienna, Austria

REFERENCES:
- [Derived] Azizzadeh M, Karimi A, Danninger K, Breyer MK, Breyer-Kohansal R, Konig A, Kaufmann CC, Boutouyrie P, Bruno RM, Mayer CC, Jager B, Hartl S, Burghuber OC, Weber T. Prevalence and determinants of vascular aging in Austria - a holistic view: the LEAD study. J Hypertens. 2025 Dec 30. doi: 10.1097/HJH.0000000000004227. Online ahead of print. PMID 41537373
- [Derived] Dal Grande A, Van Herck M, Breyer-Kohansal R, Mraz T, Karimi A, Azizzadeh M, Hartl S, Burghuber OC, Wouters EFM, Kautzky-Willer A, Schiffers C, Breyer MK. Incidence of Prediabetes and Diabetes in a European Longitudinal General Population Cohort and Its Associated Factors-Results From the Austrian LEAD Study. J Diabetes Res. 2025 Apr 22;2025:5540276. doi: 10.1155/jdr/5540276. eCollection 2025. PMID 40309217
- [Derived] Kolli F, Breyer MK, Hartl S, Burghuber O, Wouters EFM, Sigsgaard T, Pohl W, Kohlbock G, Breyer-Kohansal R. Aero-Allergen Sensitization in the General Population: Longitudinal Analyses of the LEAD (Lung Heart Social Body) Study. J Asthma Allergy. 2022 Apr 11;15:461-473. doi: 10.2147/JAA.S349614. eCollection 2022. PMID 35431559
- [Derived] Breyer-Kohansal R, Hartl S, Burghuber OC, Urban M, Schrott A, Agusti A, Sigsgaard T, Vogelmeier C, Wouters E, Studnicka M, Breyer MK. The LEAD (Lung, Heart, Social, Body) Study: Objectives, Methodology, and External Validity of the Population-Based Cohort Study. J Epidemiol. 2019 Aug 5;29(8):315-324. doi: 10.2188/jea.JE20180039. Epub 2018 Oct 20. PMID 30344197
- See also: Homepage of the Austrian LEAD Study for participants and researchers — http://www.leadstudy.at
- See also: Link to the Study profile; published in 2019 — https://www.jstage.jst.go.jp/article/jea/advpub/0/advpub_JE20180039/_pdf/-char/en
- See also: Homepage of Ludwig Bultzmann Institute for lung health — http://lunghealth.lbg.ac.at/?lang=en

RESULTS

PARTICIPANT FLOW:
Groups:
- General Population: Due to the observational, non interventional design of this study, there is only one Arm/Group (general population).
  All participants of the study receive the same measurements and quetionnaires and are re-evaluated every 4 years.
  Measurements include 1. lung function testing (spirometry/bodyplethysmography pre and post BD), 2. body composition testing (DXA Scan), 3. cardiovadcular testing (pulse wave velocity, ecg), 4. Skin Prick Test. For more detailed information please see study profile.
Period: Overall Study
Arm/Group | General Population
Started | 14966
Completed (Ongoing longitudinal study) | 14966
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Reference Population: No Intervention; obersvation healthy group (no symptoms and no lung function impairment)
Arm/Group | Reference Population
Number analyzed (Participants) | 14966
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3182
  Between 18 and 65 years | 9652
  >=65 years | 2132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8006
  Male | 6960
Region of Enrollment [Number; unit: participants]
  Austria | 14966

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Lung Function in the General Population
Description: Prebronchodilation (pre-BD) and post-BD forced spirometry measurements were determined according to international recommendations (ERS Global Lung Function Initiative). Abnromal lung function determined as forced expiratory volume in 1 second (FEV1) < Lower Limit of Normal (LLN) or forced vital capacity (FVC) < LLN or FEV1/FVC < LLN.
Time Frame: 4 years
Population: General population cohort
Measure: Count of Participants; unit: Participants
Groups:
- General Population (6-15 Years): participants at age category of 6-<15 years
- General Population (15-30 Years): participants at age category of 15-<30 years
- General Population (30-45 Years): participants at age category of 30-<45 years
- General Population (45-60 Years): participants at age category of 45-<60 years
- General Population (60-82 Years): participants at age category of 60-82 years
Arm/Group | General Population (6-15 Years) | General Population (15-30 Years) | General Population (30-45 Years) | General Population (45-60 Years) | General Population (60-82 Years)
Number analyzed (Participants) | 981 | 2012 | 2404 | 3010 | 2972
Participants
  percentage of participants with FEV1< lower limit of normal (LLN) | 65 | 145 | 178 | 226 | 252
  percentage of participants with FVC< lower limit of normal (LLN) | 52 | 121 | 96 | 108 | 143
  percentage of participants with FEV1/FVC< lower limit of normal (LLN) | 44 | 133 | 211 | 259 | 235

ADVERSE EVENTS:
Time Frame: As the LEAD study is an observational cohort study, there is no intervention, and therefore, "All-Cause Mortality", "Serious Adverse Events", and "Other (Not Including Serious) Adverse Events" were not monitored/assessed.
Description: As the LEAD study is an observational cohort study, there is no intervention, and therefore, "All-Cause Mortality", "Serious Adverse Events", and "Other (Not Including Serious) Adverse Events" were not monitored/assessed.
Groups:
- General Population: As the LEAD study is an observational cohort study, there is no intervention, and therefore no adverse effects are assessed or monitored.
Arm/Group | General Population
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes